CLINICAL TRIAL: NCT06668493
Title: A Phase 1/2, Single-arm, Open-Label Trial to Evaluate the Safety and Efficacy of Nadofaragene Firadenovec Instilled to the Renal Pelvis in Adult Subjects With Low-grade Upper Tract Urothelial Carcinoma (LG-UTUC)
Brief Title: Low-grade UTUC Treated With Nadofaragene Firadenovec Administered to Renal Pelvis
Acronym: LUNAR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000425; U1111-1292-0846 (Other: World Health Organisation (WHO))
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-07

CONDITIONS: Low-grade Upper Tract Urothelial Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Nadofaragene Firadenovec

INTERVENTIONS:
Drug: Nadofaragene Firadenovec — Repeat dose trial to investigate the safety and efficacy of nadofaragene firadenovec instilled into the renal pelvis
  Other Names: Adstiladrin

SUMMARY:
The primary purpose of this trial is to evaluate the safety & tolerability of Nadofaragene Firadenovec in subjects with LG-UTUC. To help with this evaluation, a safety lead-in period will be conducted for the first 6 subjects. Complete response is at 3 or 6 months defined as absence of any UTUC in the renal pelvis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years at the time of signing informed consent.
2. Able to give written informed consent.
3. Have biopsy-proven low-grade upper tract urothelial cancer (LG-UTUC) confirmed by a pathology report ≤2 months prior to enrolment.
4. Have ≥1 measurable papillary low-grade tumour (5-15 mm in maximum diameter), evaluated visually above the ureteropelvic junction before enrolment.

   * Subjects with low-grade tumour larger than 15 mm will be eligible if endoscopic downsizing of the tumour to 5-15 mm in maximum diameter has been performed before enrolment.
5. Willing to be available for at least 18 months after first dosing.
6. Have life expectancy >2 years, in the opinion of the investigator.
7. Have an Eastern Cooperative Oncology Group (ECOG) status of 2 or less.
8. Females of reproductive potential must have a negative highly sensitive urine or serum pregnancy test upon entry into this trial and be willing to use highly effective contraception during treatment with the investigational medicinal product (IMP) and for 6 months following the last dose. Otherwise, female subjects must be postmenopausal (no menstrual period for a minimum of 12 months) or surgically sterile. Highly effective methods of contraception include: combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner, and sexual abstinence.
9. Male subjects with female partners of reproductive potential must be surgically sterile or willing to use a condom in addition to effective contraception in their female partner during treatment with the IMP and for 3 months following the last dose.
10. Adequate laboratory values:

    * haemoglobin ≥10 g/dL
    * white blood cells (WBC) ≥4000/μL
    * absolute neutrophil count (ANC) ≥2000/μL
    * platelet count ≥100,000/μL
    * international normalized ratio (INR)* below institutional upper limit of normal (ULN)
    * activated partial thromboplastin time (aPTT)* below institutional ULN
    * aspartate aminotransferase (AST) ≤1.5 x ULN
    * alanine aminotransferase (ALT) ≤1.5 x ULN
    * total bilirubin ≤1.5 x ULN
    * sodium >135 mmol/L
    * potassium between 3.6 and 5.0 mmol/L
11. Have an estimated glomerular filtration rate (eGFR) ≥45 mL/min/1.73 m2 (for inclusion in the safety lead-in the eGFR must be ≥60 mL/min/1.73 m2 [see exclusion criteria #20]).

Exclusion Criteria:

1. UTUC characterised by one or more of the following:

   * High-grade cytology or high-grade histology
   * Multi-focal UTUC

     * Exception: Subjects with low-grade multi-focal tumours will be eligible if any ureteral tumours can be ablated before enrolment and if the total diameter of the multifocal tumours above the ureteropelvic junction is not exceeding 15 mm in diameter.
   * Bilateral disease

     * Exception: Subjects who have had bilateral disease are eligible (not in the safety lead-in) if one renal unit is removed or rendered disease-free by endoscopic ablation before enrolment.
2. Current or previous evidence of carcinoma in situ, of muscle invasive (muscularis propria) urothelial cancer in the urogenital tract presented at the screening visit.
3. Concomitant lower tract urothelial carcinoma and/or concomitant or prior urothelial carcinoma within the prostatic urethra.
4. History of high grade papillary urothelial cancer within 2 years prior to screening.
5. Current or prior treatment with mitomycin gel and/or any investigational drug for the treatment of UTUC.
6. Current systemic chemo- or immunotherapy for bladder cancer or any other malignancy.
7. Current or prior investigational treatment for Bacillus Calmette-Guerin (BCG) unresponsive non-muscle invasive bladder cancer (NMIBC) or any other investigational drug within 1 month prior to screening.
8. Current or prior retroperitoneal external beam radiotherapy within 5 years of screening.
9. Prior treatment with adenovirus-based drugs including use of other adenovirus vector medications, including COVID-19 vaccines, within 2 weeks before instillation.
10. Suspected and/or a medical history of hypersensitivity to nadofaragene firadenovec, interferon-α2b (IFN-α2b) and/or adenovector medications.
11. Urinary tract infection or bacterial cystitis (once satisfactorily treated, subjects can enter the trial).
12. Clinically significant and unexplained elevated liver or renal function tests at screening.
13. Women who are pregnant (highly sensitive urine or serum pregnancy test at screening) or breastfeeding.
14. Any other significant disease or other clinical findings which in the opinion of the investigator would prevent trial entry.
15. History of malignancy in any other organ system than the upper urinary tract within the past 5 years prior to screening. However, subjects with the following exceptions will be allowed inclusion in the trial:

    * Treated basal cell carcinoma or squamous cell carcinoma of the skin.
    * History of ≤pT2 upper tract urothelial carcinoma, at least 24 months after radical nephroureterectomy (RNU).
    * Cervical intraepithelial carcinoma (CIN) without evidence of invasive carcinoma.
    * Prostate cancer that is under active surveillance or urothelial cancer. All other genitourinary cancers are excluded.
16. Inability to deliver IMP to the pyelocaliceal system.
17. Previous BCG treatment during 6 months before the initiation of treatment.
18. Any immunosuppressive therapy within 3 months prior to screening.
19. Subjects who are immunocompromised or immunodeficient at screening.
20. Subjects with solitary kidney and/or an eGFR <60 mL/min/1.73 m2 (only applicable for subjects in the safety lead-in period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
The number of treatment-emergent adverse events reported by each subject during the trial. | Up to 30 months
Complete response | Up to 6 months
  defined as absence of any UTUC in the renal pelvis, i.e. negative urine cytology for high-grade urothelial carcinoma (centrally assessed), and either no suspicious lesions on ureteroscopy (investigator assessed) or a negative for-cause biopsy (centrally assessed).

SECONDARY OUTCOMES:
Occurrence of anti-adenoviral antibodies. | Up to 30 months
Occurrence of anti-interferon-α2b (IFN-α2b) antibodies. | Up to 30 months
Shedding of adenoviral vector with IFN-α2b. | Before dose and up to 15 days after dose
Systemic exposures to IFN-α2b protein. | Before dose and up to 15 days after dose
Systemic exposures to adenoviral vector with IFN-α2b. | Before dose and up to 15 days after dose
Systemic exposures to Syn3NODA. | Before dose and up to 15 days after dose
Duration of response, defined as the time from first achieved complete response to disease recurrence, disease progression (defined as any high-grade disease) or disease-specific death, whichever occurs first. | Up to 30 months
Urinary excretion of IFN-α2b protein. | Before dose and up to 15 days after dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (5):
- United States (5):
  - Mayo Clinic - Scottsdale Arizona, Scottsdale, Arizona
  - Indiana University, Indianapolis, Indiana
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania - Perelman Center for Advanced Medicine - Penn Urology, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center - Genitourinary (GU) Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No